CLINICAL TRIAL: NCT02509754
Title: Atrial Fibrillation Ablation Compared to Rate Control Strategy in Patients With Recently Diagnosed Impaired Left Ventricular Function: a Multicenter, Randomized Controlled Trial
Brief Title: Atrial Fibrillation Ablation Compared to Rate Control Strategy in Patients With Impaired Left Ventricular Function
Acronym: AFARC-LVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: Centro Cardiologico Monzino (Other); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); University of Padova (Other); Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Fiorenzo Gaita, M.D., Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FG062015TRN
Record Dates: First submitted 2015-07-22; First posted 2015-07-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Persistent Atrial Fibrillation; Congestive Heart Failure Due to Left Ventricular Systolic Dysfunction
Keywords: atrial fibrillation; congestive heart failure; catheter ablation; rate control; left ventricular function
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atrial fibrillation catheter ablation (Experimental): Atrial fibrillation (AF) catheter ablation is performed following each Center's common practice. Activated clotting time (ACT) is maintained above 350 seconds. The left atrium (LA) is accessed by transseptal puncture or through a patent foramen ovale. A multipolar catheter and an irrigated-tip ablation catheter are inserted into the LA and a 3-dimensional reconstruction of the LA and pulmonary veins (PVs) ostia is performed. The mainstay is to obtain a complete antral PVs isolation, defined by complete elimination of PVs potentials. PVs isolation may be accompanied by the creation of linear lesions (roof line, left isthmus) or ablation of complex fractioned atrial electrograms. Patients are discharged on oral anticoagulation and optimal medical therapy. Each center will evaluate patients for ICD implantation; a loop recorder may be implanted if within routine clinical practice.
  Interventions: Procedure: Atrial fibrillation catheter ablation
- Rate control arm (Experimental): Patients randomized to rate control only arm will undergo ICD implantation and optimization of the rate control therapy. In case of uncontrolled ventricular rate at 24-h ECG Holter, defined as a mean resting heart rate higher than 90 bpm, patients will receive atrioventricular (AV) node ablation and resyncronization therapy (CRT-D) implantation, performed following common practice at each Center. In case of failure or technical difficulties of the transvenous approach, epicardial screw-in or steroid-eluting passive lead is implanted via a limited thoracotomy. Transcatheter AV node ablation is performed as follows: a non-irrigated tip ablation catheter is introduced on the right side of the interatrial septum and ablation performed on the fast pathway region or the smallest His bundle signal. The goal of the procedure is AV modulation below 30 bpm or complete AV block.
  Interventions: Procedure: Rate control

INTERVENTIONS:
Procedure: Atrial fibrillation catheter ablation
  Arms: Atrial fibrillation catheter ablation
Procedure: Rate control — Composite of optimal medical therapy and device implantation
  Arms: Rate control arm

SUMMARY:
Atrial fibrillation (AF) and congestive heart failure (CHF) are two epidemics that share several physiopathological links. CHF patients present a significantly increased risk of developing AF and the related detrimental hemodynamic effects are even more relevant than in patients without CHF.

Within CHF patients rate control is the most widely used strategy to manage AF, having proved non-inferior to rhythm control strategies. However, by this strategy, the hemodynamic effects of AF persist, not contrasting the natural evolution towards progressive left ventricular (LV) function, cardiac output , and symptoms worsening. Rhythm control strategy, instead, has shown, in the general population, advantages over rate control concerning survival, quality of life and thromboembolic events. The main limitation is that antiarrhythmic therapy used to achieve this goal has several side effects, and that transcatheter AF ablation has been assessed only in modest sample size studies.

Available literature focusing on a direct comparison between two specific management strategies in patients with CHF and AF is limited to a small randomized study comparing pulmonary veins isolation to AV node ablation and biventricular PM implantation (PABA-CHF study). Additional indirect evidences may derive from meta-analyses of observational studies.

The investigators therefore designed this multicenter, randomized controlled trial aiming to assess if, in recently diagnosed (less than 6 months) and optimally treated CHF patients with impaired LV function, AF catheter ablation is effective in improving LV function and clinical functional class, potentially driving to a reduction of device implantations (ICD/CRTs).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia among the general population. Its prevalence increases with advanced age but also with the presence of structural heart disease. In particular patients suffering from congestive heart failure (CHF) with low left ventricular (LV) ejection fraction present a significantly increased risk of developing AF and its detrimental hemodynamic effects, due to the loss of atrial contraction, and fast and irregular beats, are an even more relevant compared to patients without CHF.

In CHF patients rate control is the most widely used strategy to manage AF; in fact, it has proved non-inferior to rhythm control strategies concerning survival rates . However, adequate ventricular rate is difficult to achieve; moreover, by rate control strategy, the detrimental hemodynamic effects of AF persist, leading to a further impair in LV function, cardiac output, and symptoms. This frequently leads to the fact that, despite optimal medical therapy (OMT) for at least 3 months, the patients require implantable cardioverter defibrillator (ICD), and, in case of poor rate control AV node ablation with resynchronization therapy (CRT). The latter, however, infer pacemaker (PM)-dependence, and relate to a not negligible risk of cardiac rhythm device peri-implantation and long-term complications (infections, leads failure).

On the other side rhythm control may represent an option. In the general population, in fact, recent evidences suggest an advantage over rate control concerning survival, quality of life and thromboembolic events. The main limitation, however, stands in how to achieve rhythm control: antiarrhythmic therapy has several side effects (amiodarone, in fact the only recommended drug, is thrived by frequent adverse events) and transcatheter AF ablation has been assessed only in modest sample size studies.

Available literature focusing on a comparison between different management strategies in patients with CHF and AF is limited. A small randomized study compared pulmonary veins (PVs) isolation to AV node ablation and biventricular PM implantation, showing improved 6-month outcome, defined by a composite end point of LV ejection fraction, 6-minutes walking distance and Minnesota Living with Heart Failure (MLWHF) questionnaire, in patients treated by PVs isolation. However, only 81 patients were enrolled in this short-term study, and no hard end point tested. More recently, and actually ongoing, the AATAC-AF study, is comparing amiodarone and catheter ablation in patients with chronic AF and an implantable device (biventricular PM or ICD). Also in this case, the preliminary results support an improved 24 month outcome, in terms of sinus rhythm (SR) achievement, quality of life and LV function, in patients undergoing AF ablation .

In addition to these direct comparisons, other indirect evidences support catheter ablation rhythm control . In a recent meta-analysis, PVs isolation, linear lesions and ablation of fragmented potentials in left atrium, although with a relatively high need for repeated procedures, have proven not only to be safe but also effective in improving symptoms (related to both CHF and AF), LV function and maintaining SR. In fact, in this analysis, 60% of the patients with a left ventricular function below 35% at baseline improved to a value above this limit following AF ablation.

We therefore designed this multicenter, randomized controlled trial aiming to assess if, in recently diagnosed (less than 6 months) and optimally treated CHF patients with impaired LV function, AF catheter ablation is effective in improving LV function and clinical functional class, potentially driving to a reduction of device implantations (ICD/CRTs).

The aim of the present study is to assess within patients with concomitant CHF and persistent AF whether AF ablation, compared to optimal rate control strategy, is superior in terms of LV function and clinical functional class. In addition, long-term outcome and complications will be recorded and compared.

This study is a prospective, multicenter, randomized, two-arms parallel-group trial. Randomization is performed through a 24-hour, centralized, computer system. Enrollment will occur at 5 centers in Italy. The study protocol will receive approval by the ethics review board at each institution before study enrollment, and patients will be randomized to undergo either arm of the study in an open fashion, due to the nature of the alternative procedures.

Written informed consent, including description of the procedure and risk of complications, is obtained from each patient before study inclusion.

At 3, 6 and 12 months from the index procedure a complete follow-up visit is performed for all patients in both study arms. Clinical assessment will include signs and symptoms of heart failure, NYHA functional class evaluation, quality of life assessment by MLWHF questionnaire and a 12-lead ECG. Additionally, all patients will undergo a complete transthoracic echocardiographic evaluation, including LV ejection fraction, end-diastolic and end-systolic volumes, LV diastolic function, LA volume, mitral regurgitation or stenosis grade, right ventricular diameter and systolic function (TAPSE). A 6-minute walking test will be performed aiming to reproducibly quantify the functional class of the patients at each scheduled evaluation. A 24-hour ECG Holter will be performed in all patients, to detect AF recurrences in the AF ablation arm, mean heart rate (both for patients in AF and SR) and ventricular arrhythmias burden. For patients implanted with a device, AF burden, ICD interventions and percentage of biventricular pacing will be recorded. Finally, the incidence of heart failure hospitalizations, ischemic or hemorrhagic strokes and all-cause mortality will be assessed in both groups. Additional clinical assessment will be performed in case of heart failure acute worsening.

No external source of funding will contribute to this study, and no conflict of interest has been to be declared. All data are independently collected, managed, and analyzed with a restricted-access database. The steering committee, is responsible for the design and conduct of the study and for the drafting and editing of the results. The steering committee will have full access to the final study data and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Recent (no longer than 6 months) diagnosis of congestive heart failure, defined as left ventricular ejection fraction lower or equal than 35% along with the presence of symptoms of heart failure, with a NYHA class II, III or ambulatory IV;
* Optimal medical therapy from at least 3 months (including a beta-blocker, an angiotensin-converting-enzyme (ACE) inhibitor or angiotensin-receptor blocker (ARB) and, in NYHA III and IV patients, spironolactone);
* Persistent atrial fibrillation (at least 3 months or, alternatively, a minimum of two previous episodes lasting longer than 7 days);
* Refractory to at least one, or intolerant to, antiarrhythmic drug/s;
* Must be able to provide written informed consent.

Exclusion Criteria:

* Reversible causes of atrial fibrillation or congestive heart failure;
* Permanent or long-standing persistent atrial fibrillation (lasting more than 1 year);
* Previous surgical or transcatheter AF ablation;
* Previously implanted CRT with or without concomitant AV node ablation;
* QRS duration above 150 msec or above 120 msec in the presence of complete left bundle branch block (class IIa indication for CRT implantation);
* Life expectancy of one year or less;
* High likelihood of undergoing cardiac transplantation within the next year;
* Contraindication to anticoagulant therapy;
* Documented intraatrial thrombus, tumor, or other abnormality that precludes catheter introduction and manipulation;
* Inability to perform a 6-minute walking test;
* Absence of optimal medical therapy as previously described;
* Cardiac surgery, myocardial infarction or percutaneous coronary intervention within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
composite of the improvement of left ventricular ejection fraction above 35% and concomitant NYHA class lower than II, measured as number of patients reporting both conditions at follow-up | 6 months

SECONDARY OUTCOMES:
6-minute walking test distance, meaused in metres | 3, 6 and 12 months
quality of life, assessed with Minnesota Living With Heart Failure questionnaire score | 3, 6 and 12 months
number of heart failure hospitalizations | 3, 6 and 12 months
number of ICD interventions | 3, 6 and 12 months
number of patients suffering ischemic or hemorrhagic stroke | 3, 6 and 12 months
all-cause mortality | 3, 6 and 12 months
  defined as number of patients died during follow-up
periprocedural major complications | 3 months
  composite of death, cerebrovascular accidents, cardiac tamponade, pneumothorax, phrenic nerve persistent injury, access site pseudoaneurysm/fistula/hematoma requiring drainage

REFERENCES:
- [Background] Benjamin EJ, Levy D, Vaziri SM, D'Agostino RB, Belanger AJ, Wolf PA. Independent risk factors for atrial fibrillation in a population-based cohort. The Framingham Heart Study. JAMA. 1994 Mar 16;271(11):840-4. PMID 8114238
- [Background] Savelieva I, John Camm A. Atrial fibrillation and heart failure: natural history and pharmacological treatment. Europace. 2004 Sep;5 Suppl 1:S5-19. doi: 10.1016/j.eupc.2004.07.003. PMID 15450275
- [Background] Wyse DG, Waldo AL, DiMarco JP, Domanski MJ, Rosenberg Y, Schron EB, Kellen JC, Greene HL, Mickel MC, Dalquist JE, Corley SD; Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) Investigators. A comparison of rate control and rhythm control in patients with atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1825-33. doi: 10.1056/NEJMoa021328. PMID 12466506
- [Background] Wang TJ, Larson MG, Levy D, Vasan RS, Leip EP, Wolf PA, D'Agostino RB, Murabito JM, Kannel WB, Benjamin EJ. Temporal relations of atrial fibrillation and congestive heart failure and their joint influence on mortality: the Framingham Heart Study. Circulation. 2003 Jun 17;107(23):2920-5. doi: 10.1161/01.CIR.0000072767.89944.6E. Epub 2003 May 27. PMID 12771006
- [Background] Doshi RN, Daoud EG, Fellows C, Turk K, Duran A, Hamdan MH, Pires LA; PAVE Study Group. Left ventricular-based cardiac stimulation post AV nodal ablation evaluation (the PAVE study). J Cardiovasc Electrophysiol. 2005 Nov;16(11):1160-5. doi: 10.1111/j.1540-8167.2005.50062.x. PMID 16302897
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822
- [Background] Gasparini M, Auricchio A, Regoli F, Fantoni C, Kawabata M, Galimberti P, Pini D, Ceriotti C, Gronda E, Klersy C, Fratini S, Klein HH. Four-year efficacy of cardiac resynchronization therapy on exercise tolerance and disease progression: the importance of performing atrioventricular junction ablation in patients with atrial fibrillation. J Am Coll Cardiol. 2006 Aug 15;48(4):734-43. doi: 10.1016/j.jacc.2006.03.056. Epub 2006 Jul 24. PMID 16904542
- [Background] Gasparini M, Auricchio A, Metra M, Regoli F, Fantoni C, Lamp B, Curnis A, Vogt J, Klersy C; Multicentre Longitudinal Observational Study (MILOS) Group. Long-term survival in patients undergoing cardiac resynchronization therapy: the importance of performing atrio-ventricular junction ablation in patients with permanent atrial fibrillation. Eur Heart J. 2008 Jul;29(13):1644-52. doi: 10.1093/eurheartj/ehn133. Epub 2008 Apr 4. PMID 18390869
- [Background] Ezzat VA, Lee V, Ahsan S, Chow AW, Segal O, Rowland E, Lowe MD, Lambiase PD. A systematic review of ICD complications in randomised controlled trials versus registries: is our 'real-world' data an underestimation? Open Heart. 2015 Feb 17;2(1):e000198. doi: 10.1136/openhrt-2014-000198. eCollection 2015. PMID 25745566
- [Background] Nof E, Epstein LM. Complications of cardiac implants: handling device infections. Eur Heart J. 2013 Jan;34(3):229-36. doi: 10.1093/eurheartj/ehs352. Epub 2012 Oct 22. PMID 23091204
- [Background] Kleemann T, Becker T, Doenges K, Vater M, Senges J, Schneider S, Saggau W, Weisse U, Seidl K. Annual rate of transvenous defibrillation lead defects in implantable cardioverter-defibrillators over a period of >10 years. Circulation. 2007 May 15;115(19):2474-80. doi: 10.1161/CIRCULATIONAHA.106.663807. Epub 2007 Apr 30. PMID 17470696
- [Background] Ionescu-Ittu R, Abrahamowicz M, Jackevicius CA, Essebag V, Eisenberg MJ, Wynant W, Richard H, Pilote L. Comparative effectiveness of rhythm control vs rate control drug treatment effect on mortality in patients with atrial fibrillation. Arch Intern Med. 2012 Jul 9;172(13):997-1004. doi: 10.1001/archinternmed.2012.2266. PMID 22664954
- [Background] Tsadok MA, Jackevicius CA, Essebag V, Eisenberg MJ, Rahme E, Humphries KH, Tu JV, Behlouli H, Pilote L. Rhythm versus rate control therapy and subsequent stroke or transient ischemic attack in patients with atrial fibrillation. Circulation. 2012 Dec 4;126(23):2680-7. doi: 10.1161/CIRCULATIONAHA.112.092494. Epub 2012 Nov 2. PMID 23124034
- [Background] Gaita F, Corsinovi L, Anselmino M, Raimondo C, Pianelli M, Toso E, Bergamasco L, Boffano C, Valentini MC, Cesarani F, Scaglione M. Prevalence of silent cerebral ischemia in paroxysmal and persistent atrial fibrillation and correlation with cognitive function. J Am Coll Cardiol. 2013 Nov 19;62(21):1990-1997. doi: 10.1016/j.jacc.2013.05.074. Epub 2013 Jul 10. PMID 23850917
- [Background] Corley SD, Epstein AE, DiMarco JP, Domanski MJ, Geller N, Greene HL, Josephson RA, Kellen JC, Klein RC, Krahn AD, Mickel M, Mitchell LB, Nelson JD, Rosenberg Y, Schron E, Shemanski L, Waldo AL, Wyse DG; AFFIRM Investigators. Relationships between sinus rhythm, treatment, and survival in the Atrial Fibrillation Follow-Up Investigation of Rhythm Management (AFFIRM) Study. Circulation. 2004 Mar 30;109(12):1509-13. doi: 10.1161/01.CIR.0000121736.16643.11. Epub 2004 Mar 8. PMID 15007003
- [Background] Gaita F, Caponi D, Scaglione M, Montefusco A, Corleto A, Di Monte F, Coin D, Di Donna P, Giustetto C. Long-term clinical results of 2 different ablation strategies in patients with paroxysmal and persistent atrial fibrillation. Circ Arrhythm Electrophysiol. 2008 Oct;1(4):269-75. doi: 10.1161/CIRCEP.108.774885. PMID 19808418
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Result] MacDonald MR, Connelly DT, Hawkins NM, Steedman T, Payne J, Shaw M, Denvir M, Bhagra S, Small S, Martin W, McMurray JJ, Petrie MC. Radiofrequency ablation for persistent atrial fibrillation in patients with advanced heart failure and severe left ventricular systolic dysfunction: a randomised controlled trial. Heart. 2011 May;97(9):740-7. doi: 10.1136/hrt.2010.207340. Epub 2010 Nov 4. PMID 21051458
- [Result] Jones DG, Haldar SK, Hussain W, Sharma R, Francis DP, Rahman-Haley SL, McDonagh TA, Underwood SR, Markides V, Wong T. A randomized trial to assess catheter ablation versus rate control in the management of persistent atrial fibrillation in heart failure. J Am Coll Cardiol. 2013 May 7;61(18):1894-903. doi: 10.1016/j.jacc.2013.01.069. Epub 2013 Mar 7. PMID 23500267
- [Result] Hunter RJ, Berriman TJ, Diab I, Kamdar R, Richmond L, Baker V, Goromonzi F, Sawhney V, Duncan E, Page SP, Ullah W, Unsworth B, Mayet J, Dhinoja M, Earley MJ, Sporton S, Schilling RJ. A randomized controlled trial of catheter ablation versus medical treatment of atrial fibrillation in heart failure (the CAMTAF trial). Circ Arrhythm Electrophysiol. 2014 Feb;7(1):31-8. doi: 10.1161/CIRCEP.113.000806. Epub 2014 Jan 1. PMID 24382410
- [Result] Khan MN, Jais P, Cummings J, Di Biase L, Sanders P, Martin DO, Kautzner J, Hao S, Themistoclakis S, Fanelli R, Potenza D, Massaro R, Wazni O, Schweikert R, Saliba W, Wang P, Al-Ahmad A, Beheiry S, Santarelli P, Starling RC, Dello Russo A, Pelargonio G, Brachmann J, Schibgilla V, Bonso A, Casella M, Raviele A, Haissaguerre M, Natale A; PABA-CHF Investigators. Pulmonary-vein isolation for atrial fibrillation in patients with heart failure. N Engl J Med. 2008 Oct 23;359(17):1778-85. doi: 10.1056/NEJMoa0708234. PMID 18946063
- [Result] Anselmino M, Matta M, D'Ascenzo F, Bunch TJ, Schilling RJ, Hunter RJ, Pappone C, Neumann T, Noelker G, Fiala M, Bertaglia E, Frontera A, Duncan E, Nalliah C, Jais P, Weerasooriya R, Kalman JM, Gaita F. Catheter ablation of atrial fibrillation in patients with left ventricular systolic dysfunction: a systematic review and meta-analysis. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1011-8. doi: 10.1161/CIRCEP.114.001938. Epub 2014 Sep 28. PMID 25262686